CLINICAL TRIAL: NCT00643084
Title: A Randomized Controlled Trial of Bowel-Prepped vs Non-Bowel-Prepped Laparoscopic Colorectal Surgery
Brief Title: Bowel Prep vs Non-Bowel Prep for Laparoscopic Colorectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Cadeddu, Dr. Margherita, McMaster University/St. Joseph's Heathcare Hamilton
Organization: McMaster University (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Bowel Prep
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Anastomotic Leak; Surgical Site Infection
Keywords: Colorectal; Bowel preparation; Laparoscopic surgery
MeSH Terms: conditions — Anastomotic Leak; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): patients will consume a low residue diet prior to surgery and have no routine bowel preparation
  Interventions: Procedure: low residue diet/no standard bowel preparation
- 2 (Other): standard bowel preparation
  Interventions: Procedure: standard bowel preparation

INTERVENTIONS:
Procedure: low residue diet/no standard bowel preparation — low residue diet/no standard bowel preparation
  Arms: 1
Procedure: standard bowel preparation — standard bowel preparation
  Arms: 2

SUMMARY:
Research Question: Are anastomotic leak and surgical site infection rates equivalent in patients having laparoscopic bowel resections without bowel preparation vs those having bowel preparation?

Bowel preparation is a distressing and uncomfortable procedure for patients undergoing laparoscopic colorectal surgery, and also carries some risk of morbidity due to dehydration, electrolyte inbalance and possible infectious complications. If it is found that there is no difference between those patients who have preoperative bowel preps and those who do not have them, then we can save these patients this additional distress and risk at the time of their surgery.

DETAILED DESCRIPTION:
Rationale: The question of whether a bowel prep is needed for colon resection in open surgery has been answered. However, in laparoscopic colorectal resections, it has not been prospectively investigated. Usually, reasons for still using a bowel prep in laparoscopic colon resections is that small instruments grasping the colon can tear it, and without a prep, stool spillage can result. As well, it may be difficult to manipulate a colon filled with stool, and difficult to identify lesions to be resected.

There are no previous randomized trials in the laparoscopic literature comparing laparoscopic colorectal resections with and without bowel preparations. There are a number of trials for open resections and one trial including both laparoscopic and open resections. Unfortunately this trial does not separate the data analysis for these two groups.

Primary and Secondary Outcomes: The question to be identified is whether anastomotic leaks, and surgical site infection rates are equivalent in patients having laparoscopic resections without bowel prep versus prepped patients.

Methodology: Once consent is obtained, the patients will be randomized into two groups-the study group who will eat a low residue diet prior to surgery and who will not undergo bowel preparation, or the control group who will complete the standard bowel preparation protocol. Both groups will have the scheduled surgery. All patients will be monitored for signs of anastomotic leak and surgical wound infection daily while in hospital and at routine follow up visits at 2 and 6 weeks postoperative. If these two complications are observed, standard treatment will be followed.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective laparoscopic colorectal resection for benign or malignant disease
* adults aged 18-85 years
* ASA 1-3

Exclusion Criteria:

* contraindications to laparoscopic surgery
* patients undergoing procedures that result in creation of a stoma or ileostomy or loop ileostomy
* patients with pre-operative perforation of established infection
* patients who cannot understand the directions for bowel preparation or low residue diet
* patients with GI obstructions
* patients who will not be able to attend the followup appointments

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Whether anastomotic leaks, and surgical site infection rates are equivalent in patients having laparoscopic resections without bowel prep versus prepped patients. | preop to 6 weeks postop

CONTACTS AND LOCATIONS:
Overall Officials: Margheta Cadeddu, MD, Principal Investigator — McMaster University; Mehran Anvari, PhD MBBS, Principal Investigator — McMaster University; Monali Misra, MD, Principal Investigator — McMaster University; Forough Farrokhyar, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University/St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Bucher P, Gervaz P, Soravia C, Mermillod B, Erne M, Morel P. Randomized clinical trial of mechanical bowel preparation versus no preparation before elective left-sided colorectal surgery. Br J Surg. 2005 Apr;92(4):409-14. doi: 10.1002/bjs.4900. PMID 15786427
- [Background] Zmora O, Lebedyev A, Hoffman A, Khaikin M, Munz Y, Shabtai M, Ayalon A, Rosin D. Laparoscopic colectomy without mechanical bowel preparation. Int J Colorectal Dis. 2006 Oct;21(7):683-7. doi: 10.1007/s00384-005-0044-y. Epub 2005 Oct 18. PMID 16231142